CLINICAL TRIAL: NCT01785407
Title: Using Stable Iron Isotopic Techniques and Serum Hepcidin Profiles to Optimize Iron Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: ETH Zürich (Unknown); University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EK 2012-N-44
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Iron Deficiency; Anemia; Iron Deficiency Anemia
Keywords: Iron bio availability; Hepcidin; Iron absorption
MeSH Terms: conditions — Iron Deficiencies; Anemia; Anemia, Iron-Deficiency | interventions — Iron-Dextran Complex; ferrous sulfate; Desiccation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 80 mg FeSO4 (Active Comparator)
  Interventions: Dietary Supplement: Iron Supplement (Ferrous Sulfate Dried)
- 40 mg FeSO4 (Active Comparator): 40 mg FeSO4
  Interventions: Dietary Supplement: Iron Supplement (Ferrous Sulfate Dried)
- 160 mg FeSO4 (Active Comparator)
  Interventions: Dietary Supplement: Iron Supplement (Ferrous Sulfate Dried)
- 240 mg FeSO4 (Active Comparator)
  Interventions: Dietary Supplement: Iron Supplement (Ferrous Sulfate Dried)

INTERVENTIONS:
Dietary Supplement: Iron Supplement (Ferrous Sulfate Dried) — Iron supplements of varying concentration will be administered to the four groups in the study. Iron bioavailability from the supplements will be assessed.
  Other Names: Ferrous Sulfate (dried)

SUMMARY:
Oral iron supplementation (OIS) is a widely-used strategy to treat iron deficiency anemia. However, absorption of OIS is often low and response is variable. To overcome this, large doses are given but this may reduce compliance due to gastric irritation. Thus, OIS doses should be low, while maximizing absorption. The prevailing serum hepcidin concentration (SHep) is the major determinant of iron absorption and erythrocyte iron utilization. Based on limited data in humans, SHep can be increased by a single OIS dose but the duration of the increase is uncertain: it may be in the range of 24 to 96 hr. Also, there are few data on how the increase in SHep determines the absorption of further doses of oral iron. Is there a threshold SHep at which subsequent iron absorption is sharply reduced? Better understanding of this relationship would be valuable to design more effective and safer OIS regimens.

Objectives: 1) Determine the duration and magnitude of the Fe induced Hepcidin rise form a single iron dose while determining its bioavailability and 2) Compare the bioavailability of a single dose to iron supplements consumed one after the other (two dosages).

DETAILED DESCRIPTION:
Background: Oral iron supplementation (OIS) is a widely-used strategy to treat iron deficiency anemia. However, absorption of OIS is often low and response is variable. To overcome this, large doses are given but this may reduce compliance due to gastric irritation. Thus, OIS doses should be low, while maximizing absorption. The prevailing serum hepcidin concentration (SHep) is the major determinant of iron absorption and erythrocyte iron utilization. Based on limited data in humans, SHep can be increased by a single OIS dose but the duration of the increase is uncertain: it may be in the range of 24 to 96 hr. Also, there are few data on how the increase in SHep determines the absorption of further doses of oral iron. Is there a threshold SHep at which subsequent iron absorption is sharply reduced? Better understanding of this relationship would be valuable to design more effective and safer OIS regimens.

Objectives: 1) Determine the duration and magnitude of the Fe induced Hepcidin rise form a single iron dose while determining its bioavailability and 2) Compare the bioavailability of a single dose to iron supplements consumed one after the other (two dosages). Methods/Subjects: Healthy female subjects will be screened for low iron status. Anemic subjects will be excluded from the study. Thirty two subjects will be included with serum ferritin <20 µg/L, C-reactive protein <5 mg/L and Hemoglobin >117 g/L. Subjects will be randomized in two groups and their Hepcidin (sHep) and iron status markers monitored at day 1 (baseline). Subjects will receive iron supplement dosages of 40, 80, 160 and 240 mg in either single or as two consecutive dosages with stable iron isotopes 54Fe, 57Fe, 58Fe in form of 4 mg of iron sulfate (FeSO4). Prior administration blood samples will be collected at 8:00, 12:00 and 16:00 to monitor sHep and iron status markers, these measurements will be repeated on the days of supplement administration. On the following days, sHep will be measured at 8:00 to quantify the duration of the iron induced hepcidin rise. In the second week, subjects receiving a single Fe dose on week 1 will receive two consecutive dosages and vice versa, while the same sampling scheme as in week one will be applied. On day 23, a last blood sample will be collected and iron incorporation of stable isotopic labels will be measured from the different dosages administered.

Outcome: The combined use of stable iron isotopes and a sensitive SHep assay will allow for better understanding of the iron-hepcidin relationship and this may enable design of more effective OIS regimens.

ELIGIBILITY:
Inclusion Criteria:

* BMI 17-25
* No anemia
* Low iron stores defined as Serum Ferritin < 20 micrograms/L
* No blood donation in in the last 4 months
* No intake of vitamin and mineral supplements 2 weeks prior and during the study

Exclusion Criteria:

* Chronic, metabolic, gastrointestinal diseases
* Taking medication
* Participation to clinical trials in the last 30 days.
* Previous participation to iron bio availability studies with stable isotopic labels.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Iron bio-availability from Oral Iron Supplements (%) | three weeks
  Iron bioavailability will be assessed with stable isotopic labels. The shift in the isotopic ratio in human whole blood 14 days after administration will be measured with Inductively coupled plasma mass spectrometry (ICP-MS).

SECONDARY OUTCOMES:
Hepcidin | three weeks
  Serum Hepcidin levels will be measured in participating subjects in concomitance with iron bioavailability.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, PhD, Principal Investigator — ETH Zürich
Locations (1):
- Laboratory of Human Nutrition, Zurich, Switzerland

REFERENCES:
- [Background] Zimmermann MB, Hurrell RF. Nutritional iron deficiency. Lancet. 2007 Aug 11;370(9586):511-20. doi: 10.1016/S0140-6736(07)61235-5. PMID 17693180
- [Derived] Moretti D, Goede JS, Zeder C, Jiskra M, Chatzinakou V, Tjalsma H, Melse-Boonstra A, Brittenham G, Swinkels DW, Zimmermann MB. Oral iron supplements increase hepcidin and decrease iron absorption from daily or twice-daily doses in iron-depleted young women. Blood. 2015 Oct 22;126(17):1981-9. doi: 10.1182/blood-2015-05-642223. Epub 2015 Aug 19. PMID 26289639